CLINICAL TRIAL: NCT03356795
Title: Multicenter Trial of Chimeric Antigen Receptor-Modified T Cells (CAR-T Cells) in the Treatment of Cervical Cancer
Brief Title: Intervention of CAR-T Against Cervical Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, President, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-17017
Record Dates: First submitted 2017-11-24; First posted 2017-11-29 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer; CAR-T; GD2; PSMA; Muc1; Mesothelin; HPV; solid tumor
MeSH Terms: conditions — Uterine Cervical Neoplasms; Medullary cystic kidney disease 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cervical cancer-specific CAR-T cells (Experimental): Peripheral blood mononuclear cells (PBMCs) of patients who have GD2, PSMA, Muc1 or Mesothelin positive cervical cancer will be obtained through apheresis, and T cells will be activated and modified to cervical cancer-specific CAR-T cells.
  Interventions: Biological: Cervical cancer-specific CAR-T cells

INTERVENTIONS:
Biological: Cervical cancer-specific CAR-T cells — 1 infusion, for 1x10^6~1x10^7 cells/kg via IV

SUMMARY:
The purpose of this clinical trial is to assess the feasibility, safety and efficacy of CAR T cells immunotherapy in patients who have GD2, PSMA, Muc1, Mesothelin or other markers positive cervical cancer. Another goal of the study is to learn more about the persistence and function of CAR T cells in the body.

DETAILED DESCRIPTION:
Cervical cancer is a cancer arising from the cervix. Human papillomavirus (HPV) infection causes more than 90% of cases. Other risk factors include smoking, a weak immune system, birth control pills, starting sex at a young age, and having many sexual partners, but these are less important. Worldwide, cervical cancer is both the fourth-most common cause of cancer and the fourth-most common cause of death from cancer in women. The treatment of cervical cancer consists of surgical intervention, radiation, chemotherapy and immunotherapy.

In this study, the participant's T-cells will be collected and modified. Then the modified T cells, called chimeric antigen receptor modified-T cells (CAR T) which can recognize specific molecules that are expressed on the surface of cervical cancer cells, are given back to the participant by intravenous infusion.

The purpose of this clinical trial is to assess the feasibility, safety and efficacy of CAR T cells immunotherapy in patients who have GD2, PSMA, Muc1, Mesothelin or other markers positive cervical cancer. Another goal of the study is to learn more about the persistence and function of CAR T cells in the body.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage III, IV or relapsed cervical cancer confirmed by histology and biopsy.
2. Age: ≥ 18 years and ≤ 70 years.
3. 4 weeks at least since last chemotherapy or radiotherapy and 2 weeks at least since last systemic steroid hormone and other immunosuppressive therapy.
4. Side Effects of Chemotherapy have subsided.
5. GD2, PSMA, Muc1, Mesothelin or other markers is expressed high (above 2+) in malignancy tissues by immuno-histochemical or flow cytometry.
6. Eastern Cooperative Oncology Group (ECOG) PS of 0 or 1.
7. Expected survival ≥ 12 weeks.
8. Initial hematopoietic reconstitution with

   * neutrophils (ANC) ≥ 1×10^6/L;
   * platelet (PLT) ≥ 1×10^8/L.
9. Proper renal and hepatic functions (ULN denotes "upper limit of normal range") with

   * serum creatinine ≤ 2×ULN;
   * serum bilirubin ≤ 3×ULN;
   * AST/ALT ≤ 2.5×ULN.
10. Oxygen saturation ≥ 90%.
11. Written, informed consent obtained prior to any study-specific procedures.

Exclusion Criteria:

1. Airway obstruction caused by tumor.
2. History of epilepsy or other central nervous system diseases.
3. Patients who require systemic corticosteroid or other immunosuppressive therapy.
4. History of prolonged or serious heart disease during QT.
5. history of serious cyclophosphamide toxicity.
6. Current or recent treatment (within the 28-day period prior to Day 0) with another investigational drug or previous participation in this study.
7. Inadequate liver and renal function with

   * serum creatinine > 1.5 mg/dl;
   * serum (total) bilirubin > 2.0 mg/dl;
   * AST & ALT > 3 x ULN.
8. Pregnant or lactating females.
9. Serious active infection during screening.
10. Active HIV, Hepatitis B virus (HBV), Hepatitis C virus (HCV) infection or uncontrolled infection.
11. Patients, in the opinion of investigators, may not be eligible or not able to comply with the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Safety of CART cells in patients using CTCAE version 4.0 standard to evaluate the level of adverse events | 3 months
  Physiological parameter (measuring cytokine response)

SECONDARY OUTCOMES:
Persistence and proliferation of CART cells in patients | 3 months
  The expansion and functional persistence of CART cells in the peripheral blood of patients will be measured by qPCR on Day 7, 14, 21, 28, 60 and 90 after infusion.
Anti-tumor effects | 1 year
  Objective response, such as complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) will be assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, PhD, Principal Investigator — Shenzhen Geno-Immune Medical Institute
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No